CLINICAL TRIAL: NCT00907725
Title: Follow-up With Serum BhCG Simplify Medical Abortion: A Randomized Controlled Trial
Brief Title: Does Follow-up With Serum Beta Human Chorionic Gonadotropin (BhCG) Simplify Medical Abortion?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009p000363
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Medical Abortion
Keywords: medical abortion; serum BhCG follow-up; ultrasonographic follow-up; follow-up methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): serum BhCG follow-up
  Interventions: Other: serum BhCG follow-up
- 2 (Other): ultrasonographic follow-up
  Interventions: Other: ultrasonographic follow-up

INTERVENTIONS:
Other: serum BhCG follow-up — Subjects in this arm will receive medical abortion follow-up using BhCG blood draw
  Arms: 1
Other: ultrasonographic follow-up — Subjects in this arm will receive medical abortion follow-up by ultrasound
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate if BhCG testing to determine the completion of medical abortion simplifies the medical abortion protocol. Investigators hypothesize that women randomized to ultrasonographic determination of completion of medical abortion will have MORE follow-up visits/interventions beyond standard protocol than those randomized to medical abortion follow-up with serum BhCG.

The investigators also hope to explore satisfaction with BhCG based follow-up among women seeking medical abortion. Investigators hypothesize that the majority of women who choose to follow-up with serum BhCG will be satisfied with this method of medical abortion follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing medical abortion
* Proficiency in English
* Working phone and willingness to be contacted by phone
* Agreeing to surveys regarding demographics, follow-up preferences, and satisfaction with chosen follow-up method

Exclusion Criteria:

* Concern for ectopic pregnancy or unable to document intrauterine pregnancy
* Clinical instability or signs of pelvic infection
* Medical conditions that contraindicate medical abortion
* Unwilling or unable to comply with study follow-up procedures
* Being in a situation where receiving phone calls or additional contact with research staff may endanger the privacy or safety of the subject (e.g., situations of domestic violence)
* Inability to give informed consent
* Previous participation in this study

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 376 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Receipt of any additional intervention or follow-up beyond the one routinely scheduled follow-up ultrasound or follow-up BhCG draw | 4 weeks

SECONDARY OUTCOMES:
Patient satisfaction with follow-up method | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Planned Parenthood
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dayananda I, Maurer R, Fortin J, Goldberg AB. Medical abortion follow-up with serum human chorionic gonadotropin compared with ultrasonography: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):607-613. doi: 10.1097/AOG.0b013e3182839fda. PMID 23635625